CLINICAL TRIAL: NCT01375634
Title: Nasogastric Tube Insertion Using Midazolam in the Emergency Department
Acronym: NIMED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Kalev Freeman, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CHRMS:M11-131-NIMED
Record Dates: First submitted 2011-06-03; First posted 2011-06-17 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Intubation; Difficult
Keywords: Intubation; Gastrointestinal
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Midazolam
- Midazolam (Experimental): Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — 2 mg intravenous over 2 minutes For patients >60 years of age or with history of pulmonary disease, 1 mg intravenous over 2 minutes
  Other Names: Versed

SUMMARY:
Nasogastric tube placement involves insertion of a flexible tube through the nose into the stomach. Placement of the tube can irritate the nose and palate and trigger gagging, causing discomfort, even if topical or local anesthetics are used. This study aims to determine if administration of an ultra-short acting sedative agent (midazolam) into a vein before the procedure, in addition to topical local anesthetic, will decrease the level of discomfort.

DETAILED DESCRIPTION:
Our overall objective is to improve patient satisfaction with nasogastric (NG) tube placement (placement of a flexible tube through the nose into the stomach) in the emergency department. Placement of an NG tube into the stomach is often performed in the emergency department (ED) setting to evacuate air, blood, or other contents. Generally performed by nursing staff at the bedside in the emergency department, the procedure may produce significant pain and discomfort for the patient despite typical measures including local medications to constrict and numb the nasal mucosa. In one questionnaire of emergency department patients at a large university hospital, placement of an NG tube was reported to be the most painful procedure, ahead of fracture reduction, abscess drainage, and urethral catheterization (Singer et al. 1999). The typical medication used for placement of an NG tube placement is administration of local, topical medications; the use of intravenous drugs to improve patient tolerance of the procedure varies widely in clinical practice (Juhl and Conners 2005). Midazolam (Versed) is an FDA-approved agent for procedural sedation, which has been used frequently at this institution for the placement of NG tubes in the emergency department. In our experience, it facilitates placement by relaxing muscles, thereby decreasing gag, and its anxiolytic and amnestic properties improve patient satisfaction. However, there are no published studies of midazolam for NG tube placement in the ED or any other setting.

The investigators will perform a randomized controlled trial to determine if a single 2mg unit midazolam dose administered intravenously decreases discomfort for patients undergoing nasogastric tube placement in the emergency department. Adult emergency department patients who require NG tubes will be screened and following informed consent they will be randomly assigned to receive either midazolam or saline control. Medications are provided by pharmacy. Registered nurses will perform the placement and administer medications; researcher, nurse and subject will be blinded to the treatment arm. Following the procedure, subjects will be asked to assess their level of discomfort and complete a brief researcher-assisted questionnaire about their experience. The nurse will also complete a questionnaire that addresses the difficulty of the procedure, level of success, and occurrence of unanticipated problems or adverse events. This study may provide support for a clinical practice to improve care for patients requiring NG tube placement in the ED.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* Receiving a nasogastric tube by a registered nurse at Fletcher Allen Health Care

Exclusion Criteria:

* less than 18 years old
* weight < 40 kg
* Need immediate nasogastric tube placement
* Endotracheal intubation
* Hemodynamically unstable
* Non-English speaking
* Without capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain score on the visual analog scale reported by patient | Within 30 minutes after completion of procedure
  Degree of pain reported by subject on a visual analog scale and a five point scale
Discomfort score on the visual analog scale reported by patient | Within 30 minutes after completion of procedure
  Degree of discomfort reported by subject on a visual analog scale and a five point scale

SECONDARY OUTCOMES:
Difficulty of tube placement | Within 30 minutes after completion of procedure
  Difficulty of nasogastric tube insertion as reported by RN on a five point scale
Complications | Within 30 minutes after completion of procedure
  Number of complications as evaluated by RN, including vomiting, epistaxis or other bleeding, gagging/choking, tracheal misplacement or knotting/kinking/coiling of tube.

CONTACTS AND LOCATIONS:
Overall Officials: Kalev Freeman, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care Emergency Department, Burlington, Vermont, United States

REFERENCES:
- [Background] Cullen L, Taylor D, Taylor S, Chu K. Nebulized lidocaine decreases the discomfort of nasogastric tube insertion: a randomized, double-blind trial. Ann Emerg Med. 2004 Aug;44(2):131-7. doi: 10.1016/j.annemergmed.2004.03.033. PMID 15278085
- [Background] Juhl GA, Conners GP. Emergency physicians' practices and attitudes regarding procedural anaesthesia for nasogastric tube insertion. Emerg Med J. 2005 Apr;22(4):243-5. doi: 10.1136/emj.2004.015602. PMID 15788820
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- See also: Emergency Medicine Research at UVM and FAHC — http://www.uvm.edu/medicine/freemanlab/?Page=em_research.html